CLINICAL TRIAL: NCT04907162
Title: Nociceptive Pain in Neuromuscular Disorders - Low Interventional Pilot Study to Assess Musculoskeletal Pain in Neuromuscular Disorders (NMD)
Brief Title: Musculoskeletal Nociceptive Pain in Participants With Neuromuscular Disorders
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Clinical Professor, LMU Klinikum
Other Study IDs: PainNMD Version 1
Record Dates: First submitted 2021-05-21; First posted 2021-05-28 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Pompe Disease (Late-onset); Myotonic Dystrophy Type 1 (DM1); Myotonic Dystrophy Type 2; Spinal Muscular Atrophy Type 3; Inclusion Body Myositis, Sporadic; Facioscapulohumeral Muscular Dystrophy 1; Healthy
Keywords: nociceptive pain; musculoskeletal
MeSH Terms: conditions — Glycogen Storage Disease Type II; Myotonic Dystrophy; Spinal Muscular Atrophies of Childhood; Myositis, Inclusion Body; Nociceptive Pain | interventions — Walk Test; Vital Signs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuromuscular disease (NMD) Patients: The patient has one of the following neuromuscular diagnoses:
  1. histologically (muscle biopsy) confirmed inclusion body myositis (IBM), or
  2. genetically confirmed late-onset Pompe disease (LOPD), or
  3. genetically confirmed spinal muscular atrophy type 3 (SMA3), or
  4. genetically confirmed myotonic dystrophy type 1, or
  5. genetically confirmed myotonic dystrophy type 2, or
  6. genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD).
  Interventions: Diagnostic Test: Beck depression inventory fast screen; Diagnostic Test: German Pain Inventory; Diagnostic Test: Brief Pain Inventory; Diagnostic Test: Fatigue Severity and Disability Scale (FSS); Diagnostic Test: Quick Motor Function Test; Diagnostic Test: Handheld Dynamometry (HHD); Diagnostic Test: Six-minute walk test (6MWT); Diagnostic Test: Pressure pain threshold; Diagnostic Test: Myotonometer Assessment; Diagnostic Test: Vital signs; Diagnostic Test: Borg Scale
- Healthy control: no known neuromuscular disorder
  Interventions: Diagnostic Test: Beck depression inventory fast screen; Diagnostic Test: German Pain Inventory; Diagnostic Test: Brief Pain Inventory; Diagnostic Test: Fatigue Severity and Disability Scale (FSS); Diagnostic Test: Quick Motor Function Test; Diagnostic Test: Handheld Dynamometry (HHD); Diagnostic Test: Six-minute walk test (6MWT); Diagnostic Test: Pressure pain threshold; Diagnostic Test: Myotonometer Assessment; Diagnostic Test: Vital signs; Diagnostic Test: Borg Scale

INTERVENTIONS:
Diagnostic Test: Beck depression inventory fast screen — Beck depression inventory fast screen questionnaire to detect severe depression for eligibility.
  Other Names: BDI-FS
Diagnostic Test: German Pain Inventory — German Pain Inventory questionnaire for evaluation of pain. Module A, abbreviated questions of module S (sociodemographic questions S1, S2, S3, S4, S5 and S8) and module L (quality of life) and V (therapies) will be used.
  Other Names: Deutscher Schmerzfragebogen (DSF)
Diagnostic Test: Brief Pain Inventory — Validated questionnaire for pain.
  Other Names: BPI
Diagnostic Test: Fatigue Severity and Disability Scale (FSS) — Validated questionnaire for perceived fatigue
  Other Names: FSS
Diagnostic Test: Quick Motor Function Test — An evaluator observes the performance of a patient and scores the items separately on a 5-point ordinal scale (ranging from 0 to 4). A total score is obtained by adding the scores of all items and ranges between 0 and 64 points.
  Other Names: QMFT
Diagnostic Test: Handheld Dynamometry (HHD) — To ensure a high level of objective measurement, muscle strength will also be assessed by handheld dynamometry. The following muscle groups will be tested: Arm abduction, elbow flexion, elbow extension, hip flexion, hip extension, knee extension, knee flexion, foot extension, foot flexion.
  Other Names: HHD
Diagnostic Test: Six-minute walk test (6MWT) — It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  Other Names: 6MWT
Diagnostic Test: Pressure pain threshold — For diagnosis of myofascial pain, pressure algometers are designed and conventionally used to measure deep pressure pain thresholds or tenderness resistance (Park, Kim et al. 2011), and the reliability of pressure pain thresholds according to raters or measurement frequencies has been proven to be relatively high (Chung, Um et al. 1992). The threshold is then determined as the arithmetic mean of the 3 series (in kPa). The measurement will be stopped immediately as the patient feels sensations of "burning", "stinging", "drilling" or "aching. Pressure algometry measurements will be performed on the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles.
  Other Names: PPT
Diagnostic Test: Myotonometer Assessment — Muscle stiffness, muscle tone, relaxation periods and viscoelasticity will be assessed by a myotonometer of selected muscles (non-invasive measurement). The method of measurement consists of recording damped natural oscillation of soft biological tissue in the form of an acceleration signal and the subsequent simultaneous computation of the parameters of State of Tension, Biomechanical and Viscoelastic properties. Measurements will be performed on the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles.
Diagnostic Test: Vital signs — Vital signs (blood pressure, heart rate, respiratory rate) will be measured before and after the six-Minute-Walk-Test (6MWT).
  Other Names: Vital parameters (VP)
Diagnostic Test: Borg Scale — the Borg scale will be assessed, which is a self-reported questionnaire designed to subjectively assess dyspnea and exertion during activity (Borg 1982). The Borg scale rates dyspnea on a scale of 0 to 10 incorporating nonlinear spacing of verbal descriptors of the level of intensity of dyspnea. A higher Borg score indicates more severe dyspnea. The Borg scale will be administered before starting the 6MWT (≤ 5 minutes) and after completing the 6MWT (≤ 5 minutes).

SUMMARY:
The primary aim is to characterize the prevalence, severity and quality of musculoskeletal nociceptive pain in adult patients with neuromuscular disorders (NMD). The secondary objectives are to evaluate whether severity and distribution of muscle pain is associated with muscle function, and to assess whether muscle pain is associated with alterations of muscle elasticity and muscle stiffness. Results of patients with neuromuscular disorders will be compared to age- and gender-matched healthy volunteers. Approx. 70 patients with neuromuscular disorders and 20 healthy volunteers will be enrolled, including patients with the following neuromuscular disorders: histologically confirmed inclusion body myositis (IBM), genetically confirmed late-onset Pompe disease (LOPD), genetically confirmed spinal muscular atrophy type 3 (SMA3), genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD), genetically confirmed myotonic dystrophy type 1 or type 2 (DM1, DM2). The duration of patient recruitment will be around 12 months.

DETAILED DESCRIPTION:
The explorative, cross-sectional low-interventional pilot study evaluates the prevalence, severity and quality of musculoskeletal nociceptive pain in participants with defined neuromuscular disorders (NMD). Adult participants with the following neuromuscular disorders will be included: histologically confirmed inclusion body myositis (IBM), genetically confirmed late-onset Pompe disease (LOPD), genetically confirmed spinal muscular atrophy type 3 (SMA3), genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD) and genetically confirmed myotonic dystrophy type 1 or type 2 (DM1, DM2). 20 healthy participants will be enrolled as a control group. The Beck depression inventory fast screen (BDI-FS) will be used as a screening. If there is a possibility of major depression (with a BDI ≥4), patients will be excluded from the study. So only patients with BDI-FS score ≤3 at screening will be enrolled. Patients will be asked to complete the following validated disease-related and quality-of-life questionnaires: German Pain Inventory (module A and abbreviated module S and L and V), Brief Pain Inventory (BPI) and Fatigue Severity and Disability Scale (FSS). Demographic and disease related data will be obtained. A neuromuscular examination will be conducted. A clinical evaluation of muscle strength using the MRC-Scale (Medical Research Council-Scale) will be performed on both sides deltoid muscles, biceps brachii muscles, triceps brachii muscles, hip flexors, hip extensors, quadriceps femoris muscles, foot extensor and foot flexor muscles as well as axial muscles and neck flexors and extensors. The Quick Motor Function Test (QMFT) with 16 items will be performed to assess muscle and movement functions of the participants. To ensure a high level of objective measurement, muscle strength will also be assessed by using handheld dynamometry. The following muscle groups will be tested: arm abduction, elbow flexion, elbow extension, hip flexion, hip extension, knee extension, knee flexion, foot extension, foot flexion. A six-minute-walk test (6MWT) will be performed once. Additionally, first signs of muscle pain or muscle cramps will be recorded (including the quality and intensity of pain). The Borg scale to rate dyspnea will be administered before starting the 6MWT and after completing the 6MWT. For diagnosis of myofascial pain, a Pressure Pain Threshold test by using a pressure algometer is included for the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles until the patient feels any sensation of pain. Measurement of muscle stiffness, muscle tone, relaxation periods and viscoelasticity of selected muscles will be assessed by a myotonometer. Data collected in this study will be reported using summary tables, figures, and patient data listings. Differences between the patients and the healthy volunteers will be analyzed.

ELIGIBILITY:
Inclusion Criteria

* The participant is willing and able to provide signed informed consent.
* The participant is able and willing to perform study-related assessments.
* The participant is ≥18 years of age
* The participant has one of the following diagnoses:

  * histologically confirmed inclusion body myositis (IBM), or
  * genetically confirmed late-onset Pompe disease (LOPD), or
  * genetically confirmed spinal muscular atrophy type 3 (SMA3), or
  * genetically confirmed myotonic dystrophy type 1, or
  * genetically confirmed myotonic dystrophy type 2, or
  * genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD).

Exclusion Criteria

* The participant is participating in another clinical study or using an investigational treatment.
* The participant, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
* The participant has currently a severe depression, assessed by the Beck depression inventory fast screen (BDI-FS) with a score ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 70 patients with defined NMD (see inclusion criteria) will be enrolled. For a control group, 20 healthy volunteers will be enrolled. All patients must be ≥ 18 years of age.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of musculoskeletal pain in defined neuromuscular diseases | Only at baseline visit
  The primary aim is to characterize the prevalence of musculoskeletal pain in adult patients with neuromuscular disorders (NMD).

SECONDARY OUTCOMES:
Association between musculoskeletal pain and muscle function, assessed by Medical research council (MRC) grading (0-5) | Only at baseline visit
  Assessed by Medical research council (MRC) grading (0-5)
Association between musculoskeletal pain and muscle function, assessed by quick motor function test (QMFT) | Only at baseline visit
  Assessed by quick motor function test (QMFT)
Association between musculoskeletal pain and muscle function, assessed by Pressure Pain Threshold (PPT) | Only at baseline visit
  Assessed by Pressure Pain Threshold (PPT)
Association between musculoskeletal pain and muscle function, assessed by a Myotonometer | Only at baseline visit
  Assessed by a Myotonometer (incl. relaxation time, stiffness, muscle tone, relaxation periods and viscoelasticity)
Assessment of Questionnaire: Beck depression inventory fast screen | Only at baseline visit
  Association between Depression and musculoskeletal pain
Assessment of Questionnaire: Brief Pain Inventory | Only at baseline visit
  Association between Depression and musculoskeletal pain
Assessment of Questionnaire: Fatigue Severity Scale (FSS) | Only at baseline visit
  Association between Depression and musculoskeletal pain
Characterization of musculoskeletal pain (quality and severity) assessed by the German Pain Questionnaire | Only at baseline visit
  Characterization of quality and severity of musculoskeletal pain
Characterization of musculoskeletal pain (quality and severity) assessed by the Brief Pain Inventory (BPI) | Only at baseline visit
  Characterization (quality and severity) of musculoskeletal pain

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wenninger, PD Dr. med., Principal Investigator — Neurologist
Locations (1):
- Friedrich-Baur-Institute, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No